CLINICAL TRIAL: NCT07079878
Title: The Effect of Bed Head Height During Feeding With Orogastric Catheter on Neonatal Growth Parameters and Feeding Tolerance in Preterm Newborns
Brief Title: The Effect of Bed Head Height During Feeding With Orogastric Catheter on Neonatal Growth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Duygu Sonmez Duzkaya, Principal Investigator, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2024/62
Record Dates: First submitted 2025-05-10; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Newborn Preterm
Keywords: preterm; oragastrik beslenme; beslenme; pozisyon
MeSH Terms: conditions — Premature Birth | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group with Bed Head Height 30° (Experimental): In the preterm newborn lying in the neonatal intensive care unit, the bed head height is adjusted to 30° 30 minutes before feeding and vital signs are monitored. After 30 minutes, the newborn is fed and vital signs are monitored during feeding. The vital signs are monitored again 30 minutes after feeding. While evaluating nutritional tolerance, abdominal distension, abdominal circumference measurement and vomiting are monitored. Growth parameters of the newborn are recorded on the growth monitoring form for 7 days. All data will be evaluated by the investigator and recorded on the intervention monitoring form.
  Interventions: Other: Group with Bed Head Height 30°
- Group with Bed Head Height 45° (Experimental): The head of the bed of the preterm newborn lying in the neonatal intensive care unit is adjusted to 45° 30 minutes before feeding and vital signs are monitored. After 30 minutes, the newborn is fed and vital signs are monitored during feeding. The vital signs are monitored again 30 minutes after feeding. While evaluating nutritional tolerance, abdominal distension, abdominal circumference measurement and vomiting are monitored. Growth parameters of the newborn are recorded on the growth monitoring form for 7 days. All data will be evaluated by the investigator and recorded on the intervention monitoring form.
  Interventions: Other: Group with Bed Head Height 45°
- Control Group (No Intervention): The bed head height of the preterm newborn lying in the neonatal intensive care unit is adjusted in accordance with the clinical routine (15°) and vital signs are monitored 30 minutes before feeding. After 30 minutes, the newborn is fed and vital signs are monitored during feeding. The vital signs are monitored again 30 minutes after feeding. While evaluating nutritional tolerance, abdominal distension, abdominal circumference measurement and vomiting are monitored. Growth parameters of the newborn are recorded on the growth monitoring form for 7 days. All data will be evaluated by the investigator and recorded on the intervention monitoring form.

INTERVENTIONS:
Other: Group with Bed Head Height 30° — 30 minutes before feeding, the bed head height of the preterm newborn is adjusted to 30° and vital signs are monitored. After 30 minutes, the newborn is fed and vital signs are monitored during feeding. The vital signs are monitored again 30 minutes after feeding. While evaluating nutritional tolerance, abdominal distension, abdominal circumference measurement and vomiting are monitored. Growth parameters of the newborn are recorded on the growth monitoring form for 7 days.
  Arms: Group with Bed Head Height 30°
Other: Group with Bed Head Height 45° — The bed head height of the preterm newborn is adjusted to 45° 30 minutes before feeding and vital signs are monitored. After 30 minutes, the newborn is fed and vital signs are monitored during feeding. The vital signs are monitored again 30 minutes after feeding. While evaluating nutritional tolerance, abdominal distension, abdominal circumference measurement and vomiting are monitored. Growth parameters of the newborn are recorded on the growth monitoring form for 7 days.
  Arms: Group with Bed Head Height 45°

SUMMARY:
Aim:The study was planned as a randomised controlled experimental study to determine the effect of bed head height applied during feeding with orogastric catheter on growth parameters and feeding tolerance of preterm newborns.

Method: The study was a randomised controlled experimental study. The sample of the study consisted of 96 newbornMethod: The study was a randomised controlled experimental study. The sample of the study consisted of 96 preterm newborns (control: 32, Group with 30° Bed Head Height: 32, Group with 45° Bed Head Height: 32) ). Data Collection Form was used as a data collection tool. The head of the newborns in the intervention group will be raised before the orogastric catheter is inserted, and the children in the control group will be routinely positioned. In this process, physiological parameters of newborns before and after positioning will be followed.

DETAILED DESCRIPTION:
The population of the study, which is planned as a prospective randomised controlled experimental study, will consist of preterm newborns hospitalised in the Neonatal Intensive Care Unit of Mersin City Hospital. While determining the sample size of the study, the scientific study titled 'Effects of the prone position and kangaroo care on gastric residual volume, vital signs and comfort in preterm infants' by Özdel & Sarı (2020) was taken as a basis as a result of literature reviews in order to determine the effect size sample size. As a result of the Power analysis (G*Power 3.1.9.2) performed according to Özdel & Sarı (2020) study; effect size = 0.967, 95% confidence interval, 95% power, it was calculated that a total of 87 newborns, at least 29 in each group, should be included. Considering the possibility of drop outs and confounding variables in the research process, the number in the groups was increased by 10%. The sample of the study was determined as 96 newborns in total, 32 newborns in each group. Randomisation In the study, 96 children in the sample will be randomly assigned to the control group, the 1st study group (Group with 30° Bed Head Height) and the 2nd study group (Group with 45° Bed Head Height). Random assignment will be made using a computer programme to determine the group of children (https://www.randomlists.com/team-generator).Place and Time of the Study The study will be conducted between July 2024 and March 2025 in the Neonatal Intensive Care Unit of Mersin City Hospital. Mersin City Hospital Obstetrics and Gynaecology Department has 2 Neonatal Intensive Care Units on the 2nd floor and 3rd floor. Research 2nd floor. In the Neonatal Intensive Care Unit, 2nd step and 3rd step patients are cared for. There are 30 incubators in the unit. Newborns with prematurity, congenital anomalies, respiratory distress, maternal preeclampsia, maternal diabetes mellitus, hypoglycaemia, and Exchange borderline phototherapy need are admitted to the Neonatal Intensive Care Unit.Data CollectionIn the study, preterm newborns who are fed with orogastric catheter in the Neonatal Intensive Care Unit will first be evaluated in terms of sampling criteria, and newborns who do not meet the criteria will be excluded from the study. The nurse who collects the data and assesses vital signs and nutritional tolerance will be the investigator herself (Nurse Özlem BORAK). Feeding of the newborns in all groups will be done in accordance with the 'Enteral Nutrition Protocol': Before starting the study, nurses working in the clinic will be trained in enteral nutrition in accordance with the 'Enteral Nutrition Protocol'.2: After obtaining written consent from the parent of the preterm baby to be fed with orogastric catheter, the application of feeding with orogastric catheter and what to be done during the procedure will be explained to the parent. Then, the newborn information form will be filled out.Stage 3: After the groups are determined in accordance with the randomisation table, the necessary materials are prepared in accordance with the feeding protocol. Stage 4: 30 minutes before feeding, the bed head height will be adjusted appropriately.5: The vital signs of the newborn (fever, pulse, respiration, oxygen saturation) will be measured 30 minutes before feeding.6: Feeding will be applied at a height of 15-20 cm, without applying pressure, at its own flow rate in 20 minutes. Stage 7: Vital signs (fever, pulse, respiration, oxygen saturation) will be measured during and 30 minutes after feeding. Stage 8: Abdominal distension will be evaluated before and 2 hours after feeding to assess nutritional tolerance. Abdominal circumference will be measured at the same time every day. Vomiting will be monitored after feeding.9: When evaluating growth parameters, weight monitoring, head circumference and height parameters will be evaluated. Weight will be monitored every day. Head circumference and height will be evaluated on the 1st and 7th days.

ELIGIBILITY:
Inclusion Criteria:

* The newborn should be in the 32-36th postnatal week
* The weight of the newborn should be over 1500 grams
* The newborn should be able to meet at least 75% of the protein and energy amount that he/she should take through the enteral route
* The newborn should be fed with an orogastric catheter
* The newborn should not need a mechanical ventilator
* The newborn should not have a congenital anomaly
* The parents should volunteer to participate in the study.

Exclusion Criteria:

* Neonates with NEC
* Newborns whose bedhead height cannot be provided due to any condition
* Previous findings of feeding intolerance
* Having a chest tube
* Parents not volunteering to participate in the study

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2024-07-05 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
Newborn Information Form | 1 day
  The information form was prepared by reviewing the relevant literature (Özdel, 2017). The neonatal information form includes 14 items including mode of delivery, 1st and 5th minute APGAR score, gestational age, birth weight, birth weight, birth head circumference, birth length, gender, mother's history of any disease during pregnancy, hospitalisation diagnosis, postnatal age, weight, height and head circumference at the time of assessment.This form will be used to identify the newborn. The average values will be calculated based on age (in days), weight (in kg), and height (in cm).
Newborn Monitoring Form | 1 day
  The follow-up form was prepared based on a review of the relevant literature (Özdel, 2017; Yüce 2020). In the newborn follow-up form, vital signs such as body temperature (Celsius), heart rate (beats per minute), respiratory rate (breaths per minute) and oxygen saturation (percentage) will be measured in the morning and evening for 7 days, and abdominal distension, abdominal circumference measurement (cm), and vomiting status will be assessed in terms of feeding tolerance, while parameters such as weight (in kilograms), head circumference (in cm), and height (in cm) will be assessed for growth monitoring over a 7-day period. The data obtained will be used to evaluate the babies' feeding.

CONTACTS AND LOCATIONS:
Overall Officials: Tarsus University, Principal Investigator — Tarsus University
Locations (1):
- Tarsus University, Mersin, Turkey (Türkiye)

REFERENCES:
- [Background] Özkan, H. (2016). Preterm ve Term Yenidoğanda Büyümenin Değerlendirilmesi. Klinik Tıp Pediatri Dergisi, 83-87.
- [Background] Özge Karakaya Suzan, N. Ç. (2020). Kolostrum: Özellikleri ve Prematüre Bebeğe Faydaları. Sted, 221-227
- [Background] Bozkurt, G., Sönmez Düzkaya D. (2015). Enteral Beslenme Uygulama Protokolü. Yenidoğan Protokolleri (s. 157-159). içinde İstanbul: Nobel Tıp Kitabevleri.
- [Background] Demet Terek, M. Y. (2019). Yenidoğan Bebeğin Beslenmesinde Temel Prensipler. Klinik Tıp Pediatri Dergisi, 233-244.
- [Background] Aysel Gürkan, B. G. (2013). Enteral Beslenme: Bakımda Güncel Yaklaşımlar Anadolu Hemşirelik ve Sağlık Bilimleri Dergisi, 116-122